CLINICAL TRIAL: NCT03573349
Title: Central Versus Peripheral GABA and Glutamate Biomarkers for Treatment Response During Two Infusions of Intravenous Ketamine for Treatment-Resistant Depression
Brief Title: Ketamine Associated ACC GABA and Glutamate Change and Depression Remission:
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Balwinder Singh, MD, MS, Assistant Professor of Psychiatry, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-011373
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Bipolar Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Other): Open-label, non-randomized
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — We will enroll 20 adults (aged 18-65 years) with treatment-resistant depression and will provide two i.v. ketamine infusions (0.5 mg/kg, infused over 40 minutes) and measure their depressive symptom responses. Biomarkers will be developed using blood samples from study subjects, taken prior to (predictive biomarkers), and following ketamine treatment (change biomarkers). This will be an open-label feasibility trial.

SUMMARY:
This is a feasibility study and the goal of this project is to evaluate whether peak ACC GABA and glutamate, quantified as a CSF-corrected absolute concentration percent change from baseline, is associated with clinical remission, Montgomery Asberg Depression Rating Scale (MADRS) total score of <10, to the anti-glutamatergic antidepressant ketamine.

As MRS is expensive, we also aim to study a correlation between change in peripheral metabolites (GABA and glutamate) and central GABA and glutamate levels.

DETAILED DESCRIPTION:
Aims: This feasibility study aims to better understand the neurobiology of major depression and how ketamine may therapeutically impact brain function. This research may provide important insights into the mechanism of ketamine response, thus, potentially increasing the likelihood of successful treatment interventions and decrease the number of ineffective treatments and/or risk for serious side effects.

SPECIFIC AIMS:

Utilizing novel dynamic sliding-window functional MR spectroscopy (fMRS) and liquid chromatography-mass spectrometry (LCMS), we aim to evaluate the relationship between GABA and glutamate (central-baseline to peak and peripheral-baseline to 24 hours) levels with a change in depression symptoms (baseline to 24 hours), after a single infusion of intravenous (IV) ketamine, in subjects with treatment-resistant depression (TRD).

ELIGIBILITY:
Inclusion Criteria:

For inclusion in this study, the following will be required:

* Ability to provide informed consent;
* Current psychiatric inpatient (voluntary only) or outpatient treatment;
* Male or female;
* Age 18-65 years;
* Meets diagnostic criteria for major depressive disorder/bipolar depression without psychotic features per the SCID DSM-IV-TR;
* PHQ-9 total score ≥ 15 at screening and at baseline (just prior to first acute phase ketamine infusion);
* Treatment-resistant depression (TRD), as defined by failure of at least two previous antidepressant treatments within the current depressive episode. Failed antidepressant treatments can include pharmacotherapy for depression at an adequate dose for at least 8 weeks, or an acute series of at least 6 administrations of electroconvulsive therapy (ECT) or an acute series of Transcranial magnetic stimulation (TMS);
* Ability to pass a comprehension assessment test related to effects of ketamine and trial objectives and criteria.

Exclusion Criteria: Based on ketamine's known difficulties with the induction of perceptual/psychomimetic symptoms, the exclusion criteria for this study will be as follows:

* Inability to speak English
* Patients with a BMI >40.
* Any current psychiatric diagnosis other than anxiety disorders needing concurrent antidepressant therapy
* Personality disorder being the primary diagnosis
* Diagnosis of schizophrenia, schizoaffective disorder, post-traumatic stress disorder, or active psychotic symptoms;
* Ongoing prescription of > 4 mg lorazepam equivalents (total) daily, or morning dosing of any benzodiazepine at the time of assessment;
* Medications known to affect glutamate (i.e., riluzole, carbamazepine) or GABA (zaleplon, zolpidem, zopiclone, valproate, gabapentin, pregabalin, tiagabine, and vigabatrin) are prohibited within two weeks prior to administration of study drug;
* Antidepressant Monoamine Oxidase Inhibitors (MAOIs) are prohibited two weeks prior to the administration of the study drug.
* CYP3A4 inducers carbamazepine and modafinil are prohibited within two weeks prior to administration of the study drug and at least 24 hours after the last dose of study drug.
* Currently undergoing TMS, vagal nerve stimulation, or deep brain stimulation as either an acute or maintenance treatment of depression;
* ECT in the past 12 months;
* Any active or unstable medical condition judged by the study psychiatrist as conferring too great a level of medical risk to allow inclusion in the study;
* Use of methamphetamine, cocaine, or cannabis. Abuse of stimulant(s) within the prior 12 months;
* Any current substance use disorder (excluding nicotine and caffeine). Note: Persons will be allowed to enroll in this study if their substance use is in complete (not partial) and sustained (> 1 year) remission;
* History of traumatic brain injury that resulted in loss of consciousness;
* Developmental delay, intellectual disability, or intellectual disorder;
* Clinical or self-reported diagnosis of delirium, encephalopathy, or related clinical diagnosis within the prior 12 months;
* Cognitive disorder (mild and major categories, per DSM-);
* Received ketamine treatment for depression within the prior 2 months;
* History of either poor antidepressive response to or poor tolerability of ketamine (any route of administration) when previously administered for treating symptoms of depression;
* History of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic for 6 months;
* Hepatic insufficiency (2.5 X ULN for AST or ALT) within 1 year of consent, past liver transplant recipient, and/or clinical diagnosis of cirrhosis of the liver;
* Gastroesophageal reflux disease
* A diagnosis of Complex Regional Pain Syndrome (CRPS);
* Pregnancy, or nursing;
* History of claustrophobia
* Any contraindication to MRI safety questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate percent change in the anterior cingulate cortex (ACC) GABA and Glutamate (baseline to peak) during a 40-minute IV ketamine infusion and remission (MADRS ≤9) at 24 hour | 24 hour
  Percent change in central metabolites and association with remission
To evaluate a correlation between percent change in ACC GABA and Glutamate/Glx levels (baseline to peak) with a change in MADRS (baseline to 24 hours). | 24 hour
  Change in central metabolite and association with change in depression scores

SECONDARY OUTCOMES:
To compare the percent change in peripheral GABA/Glutamate levels between remitters and non-remitters | 24 hour
  Change in peripheral metabolites and association with remission
To evaluate the correlation between percent change in peripheral GABA and glutamate levels with a change in MADRS scores. | 24 hour
  Change in peripheral metabolites and association with change in depression (MADRS) scores

CONTACTS AND LOCATIONS:
Overall Officials: Balwinder Singh, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh B, MahmoudianDehkordi S, Voort JLV, Han X, Port JD, Frye MA, Kaddurah-Daouk R; Mood Disorders Precision Medicine Consortium (MDPMC). Metabolomic signatures of intravenous racemic ketamine associated remission in treatment-resistant depression: A pilot hypothesis generating study. Psychiatry Res. 2022 Aug;314:114655. doi: 10.1016/j.psychres.2022.114655. Epub 2022 May 28. PMID 35738038
- [Background] Singh B, Port JD, Pazdernik V, Coombes BJ, Vande Voort JL, Frye MA. Racemic ketamine treatment attenuates anterior cingulate cortex GABA deficits among remitters in treatment-resistant depression: A pilot study. Psychiatry Res Neuroimaging. 2022 Mar;320:111432. doi: 10.1016/j.pscychresns.2021.111432. Epub 2021 Dec 24. No abstract available. PMID 34973601
- [Background] Singh B, Port JD, Voort JLV, Coombes BJ, Geske JR, Lanza IR, Morgan RJ, Frye MA. A preliminary study of the association of increased anterior cingulate gamma-aminobutyric acid with remission of depression after ketamine administration. Psychiatry Res. 2021 Jul;301:113953. doi: 10.1016/j.psychres.2021.113953. Epub 2021 Apr 20. PMID 33933839